CLINICAL TRIAL: NCT05637151
Title: Different Effects of Delayed Cord Clamping on Neonatal Bilirubin Levels Between Pregnant Women With Intrahepatic Cholestasis of Pregnancy and Normal Pregnant Women
Brief Title: Different Effects of Delayed Clamping on Neonatal Bilirubin Levels Between Pregnant Women With Intrahepatic Cholestasis of Pregnancy and Normal Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SAHoWMU-CR2022-07-206
Record Dates: First submitted 2022-11-28; First posted 2022-12-05 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Intrahepatic Cholestasis of Pregnancy
Keywords: Intrahepatic cholestasis during pregnancy; neonatal bilirubin; bilirubin; ICP; neonatal jaundice
MeSH Terms: conditions — Intrahepatic Cholestasis of Pregnancy; Jaundice, Neonatal

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ICC in pregnant women with ICP (Other): Immediate cord clamping group in pregnant women with intrahepatic cholestasis of pregnancy
  Interventions: Other: clamp time of umbilical
- DCC in pregnant women with ICP (Experimental): Delayed cord clamping group in pregnant women with intrahepatic cholestasis of pregnancy
  Interventions: Other: clamp time of umbilical
- ICC in normal pregnant women (Other): Immediate cord clamping group in normal pregnant women
  Interventions: Other: clamp time of umbilical
- DCC in normal pregnant women (Experimental): Delayed cord clamping group in normal pregnant women
  Interventions: Other: clamp time of umbilical

INTERVENTIONS:
Other: clamp time of umbilical — The umbilical cord was clamped immediately or late for more than 30s

SUMMARY:
Objective:The aim of this study was to investigate the relationship between delayed cord clamping and neonatal bilirubin levels in pregnant women with intrahepatic cholestasis of pregnancy.

Method:This observational prospective cohort study included a total of 200 pregnant women at 37-40 gestational weeks. Among them, 100 pregnant women with intrahepatic cholestasis of pregnancy were divided into 50 cases of immediate cord clamping group （ICC in pregnant women with ICP）and 50 cases of delayed cord clamping group（DCC in pregnant women with ICP）, and 100 normal pregnant women were also divided into 50 cases of immediate cord clamping group （ICC in normal pregnant women）and 50 cases of delayed cord clamping group（DCC in normal pregnant women）. The bilirubin levels of neonates in each group were compared.

ELIGIBILITY:
Inclusion Criteria:

1. The pregnant woman is born at a gestational age of 37-40 weeks;
2. The pregnant woman has a single child;
3. Regular obstetric examination durinv pregnancy with complete obstetric examination data was diagnosed as intrahepatic cholestasis of pregnancy(ICP).

Exclusion Criteria:

1. Pregnancy complicated with medical and surgical diseases, such as thyroiddysfunction and chronic hypertension;
2. Insufficiency of vital organ function or complicated tumor;
3. Pregnant women with other pregnancy complications besides ICP, such as preeclampsia, etc.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
the neonatal bilirubin values | 2-4 days after birth
  the neonatal bilirubin values

CONTACTS AND LOCATIONS:
Overall Officials: Ying Hua, Study Director — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- department of obstetrics of Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China